CLINICAL TRIAL: NCT06343064
Title: A Phase Ib/II Study of Vebreltinib Plus PLB1004 in EGFR-mutated, Advanced NSCLC With MET Amplification or MET Overexpression Following EGFR-TKI
Brief Title: Vebreltinib Plus PLB1004 in EGFR-mutated, Advanced NSCLC With MET Amplification or MET Overexpression Following EGFR-TKI
Acronym: KYLIN-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Avistone Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PLB1001/PLB1004-NSCLC-Ib/II-01
Record Dates: First submitted 2024-03-21; First posted 2024-04-02 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: Non-Small-Cell Lung Cancer; EGFR; NSCLC; Lung Cancer; MET Amplified; MET Expression
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Phase Ib:Vebreltinib 100mg/150mg/200mg BID + PLB1004 80mg/160mg QD (Experimental): In the dose-escalation and dose-expansion phase, patients received oral Vebreltinib 100mg/150mg/200mg BID plus PLB1004 80mg/160mg once daily.
  Interventions: Drug: Vebreltinib; Drug: PLB1004
- Phase II:Cohort 1 (Experimental): In phase II-Cohort 1:Failed first-generation or second-generation EGFR inhibitors, negative T790M mutation and c-Met amplification(GCN≥6).Patients received oral Vebreltinib（RP2D）plus PLB1004 （RP2D）.
  Interventions: Drug: Vebreltinib; Drug: PLB1004
- Phase II:Cohort 2 (Experimental): In phase II-Cohort 2 :Failed third-generation EGFR inhibitors, c-Met amplification(GCN≥6).Patients received oral Vebreltinib（RP2D）plus PLB1004 （RP2D）.
  Interventions: Drug: Vebreltinib; Drug: PLB1004
- Phase II:Cohort 3 (Experimental): In phase II-Cohort 3 :Failed first-generation or second-generation EGFR inhibitors, c-Met over expression.Patients received oral Vebreltinib（RP2D）plus PLB1004 （RP2D）.
  Interventions: Drug: Vebreltinib; Drug: PLB1004

INTERVENTIONS:
Drug: Vebreltinib — Phase Ib is a dose escalation study, the initial dose of Vebreltinib is 100mg/150mg/200mg,according to the result of Phase Ib, will confirm the RP2D.
  Other Names: Bozitinib; PLB1001
Drug: PLB1004 — Phase Ib is a dose escalation study, the initial dose of PLB1004 is 80mg/160mg,according to the result of Phase Ib, will confirm the RP2D.

SUMMARY:
Efficacy and Safety Evaluation of Vebreltinib Plus PLB1004 in EGFR TKI Relapsed MET Amplified or MET Expression in NSCLC

DETAILED DESCRIPTION:
Open label, multicenter Phase Ib/II clinical study to evaluate the safety, efficacy, and pharmacokinetics of Vebreltinib in combination with PLB1004 in patients with locally advanced or metastatic non-small cell lung cancer with MET overexpression or MET amplification following EGFR-TKI treatment failure.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign a written informed consent document.
2. Aged at least 18 years old.
3. Histologically or cytologically confirmed locally advanced or metastatic NSCLC (stage IIIB~IV).
4. EGFR mutations, including exon 19 deletion and exon 21 L858R.
5. C-Met overexpression and/or c-Met amplification confirmed after treatment with EGFR-TKI.
6. At least one measurable lesion as defined by RECIST V1.1.
7. ECOG performance status 0 to 1.

Exclusion Criteria:

1. Previous treatment with MET inhibitors or HGF-targeted therapy.
2. There are mutations of ALK or ROS1.
3. Have symptomatic and neurologically unstable central nervous system (CNS) metastases or CNS disease that requires increased steroid doses for control.
4. Pregnant or nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]). | 3 years
  In phase Ib，Incidence of Treatment-Emergent Adverse Events (TEAEs),
Incidence of dose-limiting toxicities (DLT) as defined in the protocol. | 28 days
  In phase Ib，Number of patients with at least 1 dose-limiting toxicity (DLT), which is any toxicity defined as a DLT in the Clinical Study Protocol
Overall Response Rate (ORR） | 3 years
  In phase II,ORR is defined as the proportion of subjects with confirmed best overall response of complete response (CR) or partial response (PR) according to RECIST 1.1.

SECONDARY OUTCOMES:
Pharmacokinetics of Vebreltinib and PLB1004 : Area under the concentration time curve (AUC) | From date of first dose up until 28 days post last dose
  In phase Ib，Measurement of PK parameters: Area under the concentration time curve (AUC)
Pharmacokinetics of Vebreltinib and PLB1004: Maximum plasma concentration of the study drug (C-max) | From date of first dose up until 28 days post last dose
  In phase Ib，Measurement of PK parameters: Maximum observed plasma concentration of the study drug (C-max)
Pharmacokinetics of Vebreltinib and PLB1004: Time to maximum plasma concentration of the study drug (T-max) | From date of first dose up until 28 days post last dose
  In phase Ib，Measurement of PK parameters: Time to maximum observed plasma concentration of the study drug (T-max)
Incidence of Treatment-Emergent Adverse Events | 3 years
  In phase II，Incidence of Treatment-Emergent Adverse Events (TEAEs),A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China